CLINICAL TRIAL: NCT00252096
Title: Nucleic Acid Amplification Tests for the Diagnosis of Pharyngeal and Rectal Chlamydia Trachomatis and Neisseria Gonorrhoeae Infections
Brief Title: Nucleic Acid Amplification Tests (NAATs) for the Diagnosis of Pharyngeal and Rectal Chlamydia and Gonorrhea Infections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: University of Alabama at Birmingham (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CDC-NCHSTP-3881; CA U36/CCU300430 PA05048; ASPH S2070-22/22
Record Dates: First submitted 2005-11-10; First posted 2005-11-11 (Estimated); Last update posted 2012-09-27 (Estimated); Status verified 2012-09

CONDITIONS: Chlamydia Infections; Gonorrhea
Keywords: Diagnosis; Chlamydia trachomatis; Neisseria gonorrhoeae; Nucleic acid amplification test; Rectum; Pharynx
MeSH Terms: conditions — Chlamydia Infections; Gonorrhea; Disease | interventions — Nucleic Acid Amplification Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Nucleic acid amplification test

SUMMARY:
Investigators at the University of Alabama in Birmingham in collaboration with investigators from the Centers for Disease Control in Atlanta are evaluating the performance of three commercial nucleic acid amplification tests for the detection of Chlamydia trachomatis and Neisseria gonorrhoeae in pharyngeal and rectal swab specimens. Cultures for C. trachomatis and N. gonorrhoeae are performed as additional reference tests. Study subjects are men and women attending sexually transmitted disease (STD) and HIV care clinics in Birmingham, Alabama, who report sexual behaviors that place them at risk for pharyngeal or rectal sexually transmitted infections.

DETAILED DESCRIPTION:
In the latter part of the 1990's, testing for Chlamydia trachomatis and Neisseria gonorrhoeae infections was revolutionized by the introduction of nucleic acid amplification tests (NAATs) which achieve greater sensitivity than traditional culture methods by exponentially replicating the nucleic acid of these organisms. The specimens collected for NAATs are easier to transport and NAATs permit collection of less invasive specimens for testing (i.e. voided urine or patient-collected vaginal swabs for women rather than urethral or endocervical swabs). Despite their somewhat higher costs, these tests have been found to be preferred by patients (because specimens can be collected less invasively), by clinicians (because of both their ease of collection and increased sensitivity), and to permit expanded screening both in traditional clinical settings and at outreach sites where testing has not typically been done in the past.

NAATs have been cleared by FDA for testing of genital specimens (cervical and male urethral swabs and urine), but the performance of NAATs has not been adequately evaluated for diagnosis of C. trachomatis and N. gonorrhoeae infections occurring at rectal or pharyngeal sites of sexual exposure. Increasing numbers of heterosexual individuals might be engaging in orogenital or rectal sexual activity, especially adolescents and young adults who might view such exposures as less risky with respect to pregnancy and sexually transmitted diseases (STD) than penile-vaginal intercourse. Pharyngeal and rectal exposures, often without use of condoms, are relatively common among MSM. Recent demonstration of resurgent sexually transmitted diseases and unsafe sexual practices among men-who-have-sex-with-men (MSM), including those who are infected with the human immunodeficiency virus (HIV), provides an especially strong public health imperative to the need for careful evaluation of NAATs with pharyngeal and rectal specimens.

The primary aim of this study is to compare the performance of the three NAATs that are available commercially to test pharyngeal and rectal specimens for C. trachomatis and N. gonorrhoeae infections with culture, the current method of choice, and with each other. In order to enroll adequate numbers of individuals with such infections, the study will be conducted during a 3-year period in a STD clinic and two HIV care clinics located in Birmingham, AL. Enrollment will be confined to individuals who are at high risk for genital C. trachomatis or N. gonorrhoeae infection, or who give a history of orogenital or rectal sexual exposures. An effort will be made to balance enrollment of heterosexual individuals and MSM, but resource limitations require that sample sizes be based on combining these subgroups.

No adequate criterion-standard for pharyngeal or rectal infections exists due to the probable, but poorly defined, low sensitivity of the current standard, culture. Fortunately, the 3 NAATs employ different C. trachomatis and N. gonorrhoeae molecular targets and methods of nucleic acid amplification. By including all 3 NAATs plus culture in the study, combinations of the results of culture and a NAAT or of two NAATs can be utilized to take advantage of the likely independence of testing errors among truly uninfected subjects to construct more satisfactory criterion standards for infection for the purpose of estimating and comparing their sensitivities and specificities. A secondary aim of the study will be to compare this methodological approach, utilizing a traditional statistical and clinical epidemiological approach, with alternative methods that have been more widely used but strongly criticized by statisticians and clinical epidemiologists and with newer methods designed to meet these criticisms and to be more efficient than the traditional statistical approaches.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 15 years.
* If male, history of fellatio, cunnilingus, or receptive anal sex within the last two months.
* If female, presenting for treatment of N. gonorrhoeae and/or C. trachomatis or contact to N. gonorrhoeae, C. trachomatis, or nongonococcal urethritis.
* If female, history of fellatio or history of anal sex within the last two months.

Exclusion Criteria:

* Declines to participate.
* History of receipt of antimicrobial agents active against N. gonorrhoeae or C. trachomatis in the preceding 30 days.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3900 (Estimated)
Dates: Start 2003-06; Primary Completion 2006-01 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Detection of Chlamydia trachomatis or Neisseria gonorrhoeae infections

CONTACTS AND LOCATIONS:
Overall Officials: Laura H. Bachmann, MD, MPH, Principal Investigator — University of Alabama at Birmingham; Edward W. Hook, III, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States